CLINICAL TRIAL: NCT03708952
Title: Lifestyle and Dietary Pattern in Relation to Precursor Lesions of Colorectal Cancer and Cardiometabolic Diseases Among High-risk Populations in Lanxi, China
Brief Title: Lifestyle and Dietary Pattern in Relation to Precursor Lesions of Colorectal Cancer and Cardiometabolic Diseases
Status: Active, not recruiting | Type: Observational
Sponsor: Zhejiang University (Other)
Collaborators: Lanxi Hospital of Traditional Chinese Medicine (Other); Lanxi Red Cross Hospital (Unknown)
Responsible Party: Principal Investigator, Jingjing Jiao, Associate Professor, Zhejiang University
Other Study IDs: cohort- colorectal cancer
Record Dates: First submitted 2018-10-14; First posted 2018-10-17 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Polyps; Cardiovascular Diseases
Keywords: Dietary factors; Precursor lesions of colorectal cancer; Lifestyle; Polyps; Cardiovascular Diseases
MeSH Terms: conditions — Polyps; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The investigators collect blood samples.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The association between lifestyle and dietary patterns with precursor lesions of colorectal cancer and cardiometabolic diseases is still unclear. This study is conducted in Jinhua, a city with a high prevalence of colorectal cancer in China, to assess the relationship between lifestyle and dietary factors with precursor lesions of colorectal cancer and cardiometabolic diseases.

DETAILED DESCRIPTION:
Investigations of lifestyle and dietary factors in relation to precursor lesions of colorectal cancer and cardiometabolic diseases are limited in China. The investigators aim to collect the basic characteristics of participants at baseline, including sex, age, smoking, exercise, marriage, education level, dietary factors and so on, to assess the associations between lifestyle and dietary factors with precursor lesions of colorectal cancer and cardiometabolic diseases. This large cohort - the Lanxi Pre-colorectal Cancer Cohort (LP3C) also included several subcohorts consisting of patients with CVD, diabetes, hypertension, metabolic syndrome, obese/overweight or fatty liver disease. Results from this study will be valuable for colorectal cancer and cardiometabolic disease prevention in China.

ELIGIBILITY:
Inclusion Criteria:

* Subject aged ≥45 and ≤74 years old
* Subject has complete data on diet and follow-up time

Exclusion Criteria:

* Colorectal cancer
* Severe intestines problems

Ages: 45 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects are eligible residents from 16 towns and villages of Jinhua, China.
Sampling Method: Probability Sample
Enrollment: 25000 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Numbers of participants with polyps | From entry into the study (baseline:2018-2022) until 2028
  All polyps

SECONDARY OUTCOMES:
Numbers of participants with different subtypes of polyps | From entry into the study (baseline:2018-2022) until 2028
  Subtypes of polyps, including serrated polyps, hyperplastic polyps, sessile serrated polyps/adenoma
Numbers of participants with cardiometabolic diseases | From entry into the study (baseline:2018-2022) until 2028
  Cardiometabolic diseases including cardiovascular disease, diabetes, and hypertension

OTHER OUTCOMES:
Numbers of participants died | From entry into the study (baseline:2018-2022) until 2028
  All-cause and cause-specific mortality outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Weifang Zheng, MD, Principal Investigator — Lanxi Red Cross Hospital; Jingjing Jiao, Principal Investigator — Zhejiang University; Pan Zhuang, Principal Investigator — Zhejiang University
Locations (2):
- China (2):
  - Lanxi Hospital of Traditional Chinese Medicine, Jinhua, Zhejiang
  - Lanxi Red Cross Hospital, Lanxi, Zhejiang